CLINICAL TRIAL: NCT06353308
Title: Effectiveness of an Online Intervention Using a Feminist Approach on Gender Equality Promotion and Sexual Violence Prevention in China: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of an Online Intervention Using a Feminist Approach on Gender Equality Promotion and Sexual Violence Prevention in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA230308
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Sexual Violence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Sexual Health intervention (Placebo Comparator): Participants will receive their general online sexual health education programming.
  Interventions: Behavioral: Sexual health intervention
- Feminist Sexual Health Intervention (Experimental): Participants will receive online feminist sexual health program.
  Interventions: Behavioral: Sexual Violence Prevention

INTERVENTIONS:
Behavioral: Sexual Violence Prevention — The intervention included a game, five short videos, two posters, and five online quizzes, which were provided with a frequency of two posts per week and a final real-time online workshop. Materials included content on the spectrum of gender and sexual identities and orientations, gender and sexual roles, consent and communication, body positivity and self-acceptance, sexual pleasure and desire, as well as risky sexual behavior associated with dating app use and the legal issues and risks of sexual assault, such as precautionary steps and available resources.
  Arms: Feminist Sexual Health Intervention
Behavioral: Sexual health intervention — This general online sexual health education consisted of online videos, quizzes and game that covered a wide range of diverse topics on love, sex and relationships such as healthy and respectful relationships, body self-esteem, sexual identity and orientation, sexual rights and decision making, in addition to the conventional focus on sexual dysfunction and disease aversion.
  Arms: General Sexual Health intervention

SUMMARY:
This paper presents the findings of a clustered randomized controlled trial (cRCT) that evaluated the effectiveness of an online feminist sexual health intervention among Chinese young adults, providing insights into the impacts of this innovative approach and contribute to the growing body of literature on feminist interventions for sexual health and equality promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Young adults aged between 18-29 years old who possessed a mobile phone
2. Had prior experience in using social media
3. Were able to read and understand Chinese

Exclusion Criteria:

1. Those with a physical impediment (e.g., blindness) preventing them from accessing the mobile content

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Rape myth acceptance | From enrollment to the end of treatment at one week and three months
  Illinois Rape Myth Acceptance Scale -Short Form, which consists of 17 items (1=not at all agree, 7=very much agree) assessing respondents' belief in rape myths (e.g., "Rape happens when a man's sex drive gets out of control"). The scores range from 17 to 119, with lower scores indicating less subscription to rape myths.

SECONDARY OUTCOMES:
Sociocultural Attitudes toward Appearance | From enrollment to the end of treatment at one week and three months
  Sociocultural Attitudes toward Appearance Questionnaire-3 consisted of eight items assessing the degree to which an individual accepts and internalizes societal standards of beauty. Examples include "I tend to compare my body to people in magazines and on TV" and "Women who appear in TV shows and movies project the type of appearance that I see as my goal." Each item is rated on a five-point Likert scale. The scores range from 8 to 40, with lower scores indicating less endorsement of sociocultural beauty standards.
Sexual Attitudes Scale | From enrollment to the end of treatment at one week and three months
  Sexual Attitudes Scale is a 22-item scale that includes: Permissiveness (six items); Responsibility (four items); Pleasure (four items); Instrumentality (four items); and Communion (four items). The factor items were rated on a five-point Likert-type scale ranging from 1 (strongly agree) to 5 (strongly disagree). After reverse-coding the negatively worded items, the item scores of each factor are summarized to obtain a total score for the factor. High scores indicated a high level of acceptance of the factor. The scores range from 22 to 110.
Sexual Desire Inventory | From enrollment to the end of treatment at one week and three months
  Sexual Desire Inventory is a self-reported scale developed to assess sexual desire. It has 14 items in two aspects: Dyadic Sexual Desire (DSD)and Solitary Sexual Desire (SSD). Items1,2,10 and14 are rated on 8-point scales with responses from 0 (Not at all or Always) to 7 (> once a day or < one day) and Items 3-9, 11-13 are rated on 9-point scales with responses from 0 (No desire, Not important at all, or Extremely low desire) to 8 (Strong desire, Extremely important, or High desire). High scores indicated a high level of sexual desire. The scores range from 0 to 108.

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Hong Kong, Hong Kong, Hong Kong